CLINICAL TRIAL: NCT04549961
Title: 123 nutritionDay in Worldwide ICUs: An International Audit and Registry on Nutrition and Outcome.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Collaborators: European Society for Clinical Nutrition and Metabolism (Other); Austrian Society for Clinical Nutrition (Other)
Responsible Party: Principal Investigator, Michael J. Hiesmayr, Professor of Anesthesia and Intensive Care, Medical University of Vienna
Other Study IDs: 509/2006 (ICU)
Record Dates: First submitted 2020-08-06; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition | interventions — Nutritional Status; Food Service, Hospital; Dietary Supplements; Enteral Nutrition; Parenteral Nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- patients admitted to intensive care units: all patients that are present on an intensive care unit on nutritionday
  Interventions: Other: Nutrition

INTERVENTIONS:
Other: Nutrition — type and amount of food eaten or type and amount of oral nutritional supplements as well as enteral or parenteral nutrition
  Other Names: hospital food; oral nutritional supplements; enteral nutrition; parenteral nutrition

SUMMARY:
The aim of this project is to increase knowledge and awareness about nutrition of ICU patients among the staff by evaluating nutrition care on an international level. In order to be able to facilitate bench-marking of ICU's with a national and international standard and actual best practice, we intend to provide a multi-lingual data acquisition tool to determine actual nutrition care in an ICU's.

nutritionDay in Worldwide ICUs is a one day international cross-sectional audit.

DETAILED DESCRIPTION:
One day international cross-sectional audit in all types of intensive care units. Data are collected with the help of questionnaires. Anonymised data entry into the audit database is done with individual and anonymous center and unit-codes.

There are 4 questionnaires to be completed on nutritionDay.

1. Unit Sheet: asks for nutrition related organisational and structural information on the ward.
2. Patient Medical Information Admission Day: asks for patients status (gender/age/weight/height etc.), date of ICU admission and laboratory parameters on admission day.
3. Patient Medical Information Actual Day: includes questions about treatment (insulin therapy/antibiotic treatment, etc.) and laboratory parameters on actual day.
4. Patient Nutrition: comprises questions about enteral and parenteral nutrition. Number of days of parenteral/enteral feeding, planned amount of calories per day and the patients well being.

Outcome Evaluation: re-assesses the patient's outcome 60 days after nutritionDay (discharged, still in hospital, transferred, death...).

Participation rules:

A user needs to register to nutritionDay as a member to the nutritionDay network. Each may choose a personal user name. Each user needs to provide a valid email address. After responding to a validation email the user is registered with the chosen user name. User details are stored on a system that is not connected to the nutritionDay registry at any time. One user may serve as contact for several units and centers.

A user may order codes for participation for one or several centers and units. Access to the registry is only possible with a center code and unit code. These codes are selected from a list of random numbers.

Audit/registry recruitment plan:

Participation to the registry is voluntary. There is actually no participation fee. All necessary information can be obtained from a dedicated website (www.nutritionday.org). Participation can be promoted via international and national scientific societies, universities, health care organisations or governmental agencies as well as via advertisement at international and national congresses. The target would be intensive care units within hospitals of different sizes and level of care.

Risk and benefit assessment:

The benefit for each patient is that awareness and knowledge about nutrition related factors and treatment options in the treating unit is increased. There is no individual risk since the audit is purely observational.

The benefit for the individual unit is to receive an extensive benchmarking report displaying the unit data in comparison with all units from the same specialty from the previous 3 years immediately after the end of data entry and a validation step. Units or groups of units may request specific reports that can be obtained only after a case by case agreement and financial coverage. All data used as a reference for benchmarking purpose are from units where a minimum of 60% of actually present patients have been recruited and the outcome at day 60 is available in more than 80% of these patients. There is no risk for the unit since anonymity of unit is structurally strictly maintained.

The benefit for the registry up-to-date data enabling benchmarking in pace with medical and care evolution. Moreover the registry data are used for research of the scientific community.

Data security:

On the datasheets the unit and the hospital/center are identified by a numeric code delivered after application to the nutritionDay coordinating center by an automatic system. The only requirement is a valid email address for direct communication with the unit.

Patients are usually identified on the locally used questionnaires by initials and age, but use of initials is not mandatory. Consecutive numbering is also possible. Only the participating unit has to trace patients identifier to be able to collect hospital outcome at day 60 after nutritionDay and to answer automatic requests for data clarification during the data quality feedback.

During data entry into the electronic registry only anonymous codes for center, unit and patients are possible. Thus the data handling centre cannot trace data back to an individual patient. The access to data entry is protected by anonymous center-code and unit-code.

Typically all data are collected via a dedicated website accessed via www.nutritionday.org .

The protected data server is run by the Center for Medical Statistics Informatics and Intelligent Systems (CEMSIS) of the Medical University Vienna. The data server is mirrored and backed up. The data server is protected within the University Firewall against external access.

Data feedback and individual unit report

All participating units are entitled to receive a bench-marking report from the registry. The report generator is started by the participating unit, when data entry has been completed. As a first step each unit receives a data feedback sheet that is based on an electronic data plausibility and missing data analysis. After stating that all data are correctly entered the final report can be generated. This final report offers complete descriptive statistics of the unit data compared to the reference data from the previous 4 years of the corresponding specialty. Only data from units fulfilling a high data quality standard are used for the reference. More than 60% of the patients present in the unit need to participate and 80% of these patients need to have their outcome recorded. Optionally the period used for comparison can be extended until 2007. All descriptive statistics represent prevalent data and are not corrected for cross-sectional sampling to allow direct data control and interpretation.

All downloaded reports of a unit are consecutively numbered and stored for documentation purpose.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to an intensive care unit on nutritionDay
* patients aged 6 and older

Exclusion Criteria:

* refusal of patient or relatives to participate in nutritionDay
* patient aged 5 and under

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted to an intensive care unit on nutritionDay.
Sampling Method: Non-Probability Sample
Enrollment: 35000 (Estimated)
Dates: Start 2007-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
60 day hospital mortality | 60 days
  death within 60 days of sampling day
Length of ICU stay | 60 days
  difference in days between ICU admission and ICU discharge
Route of nutrition | at nutritionDay (the sampling day)
  artificial nutrition is defined in 4 categories (yes/no):
  1. enteral nutrition: nutrition provided via a tube into the gastro-intestinal tract
  2. parenteral nutritoin: nutrition infused via a vascular access to a peripheral or central vein
  3. oral nutrition: any nutrition taken by mouth either as food or as oral nutritional supplement
  4. no nutrition: no provision of nutrients via enteral, parenteral or oral route
planned and delivered amount of nutrition | 24 hour period before nutritionDay and 24 hour period of nutritionDay (the sampling day)
  amount of nutrition in kilocalories from all routes:
  1. planned amount
  2. delivered amount
  3. planned amount for the next day

SECONDARY OUTCOMES:
Structural parameters: number of ICU beds | baseline ( on the day of cross-sectional data collection nutritionDay)
  number of staffed ICU beds
Structural parameter: human resources | baseline ( on the day of cross-sectional data collection nutritionDay)
  number of physician, nurses, dietician present in the ICU during the morning shift

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Hiesmayr, MD, MSc, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University Vienna, CEMSIIS, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
Upon submission of a research proposal anonymised data are shared with researcher. Each proposal is submitted to the supervisory board for approval.
Supporting Information: Study Protocol, ICF
Time Frame: 2 months
Access Criteria: submit a research proposal, acceptance by the nutritionDay scientific committee and signature of a data sharing contract according to the legal department of medical University Vienna.

REFERENCES:
- [Background] Bendavid I, Singer P, Theilla M, Themessl-Huber M, Sulz I, Mouhieddine M, Schuh C, Mora B, Hiesmayr M. NutritionDay ICU: A 7 year worldwide prevalence study of nutrition practice in intensive care. Clin Nutr. 2017 Aug;36(4):1122-1129. doi: 10.1016/j.clnu.2016.07.012. Epub 2016 Aug 9. PMID 27637833
- See also: nutritionDay project website — http://www.nutritionday.org